CLINICAL TRIAL: NCT02417584
Title: The Role of Compliance With Positive Airway Pressure Use on Blood Pressure in Patients With Obstructive Sleep Apnea
Brief Title: Efficacy of PAP Therapy on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, MD, PhD, Consultant at NHS, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAPBP-01
Record Dates: First submitted 2015-04-11; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Obstructive Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- positive airway pressure (PAP) (Experimental): Treatment with positive airway pressure (PAP)
  Interventions: Device: positive airway pressure (PAP)

INTERVENTIONS:
Device: positive airway pressure (PAP) — Positive Airway Pressure (PAP) is a non-invasive machine providing air pressure f to prevent the collapse of the oropharyngeal walls and the obstruction of airflow during sleep, which occurs in obstructive sleep apnea hypopnea syndrome.

SUMMARY:
The aim of the study was to determine the long term effects of compliance with positive airway pressure therapy on blood pressure in both hypertensive and normotensive patients with obstructive sleep apnoea hypopnoea syndrome.

DETAILED DESCRIPTION:
Scientific data about the causal role of obstructive sleep apnoea hypopnoea syndrome (OSAHS) in the development of systemic hypertension and the effects of positive airway pressure (PAP) treatment on blood pressure (BP) control are continuously increasing; however they are controversial. We aimed to determine the long term effects of compliance with PAP therapy on BP in both hypertensive and normotensive patients with OSAHS.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed OSAHS by polysomnography according to standard criteria
* no history of previous PAP therapy
* normotensive and hypertensive patients
* an above-elementary school education.

Exclusion Criteria:

* refusal to participate
* refusal of PAP therapy
* secondary hypertension
* central sleep apnea syndromes
* obesity hypoventilation syndrome
* restrictive ventilator syndromes
* history of established cardiovascular disease
* severe congestive heart failure
* a history of life-threatening arrhythmias
* severe cardiomyopathy
* significant chronic kidney disease
* long-term oxygen therapy
* family or personal history of mental illness
* drug or alcohol abuse
* severe cognitive impairment
* concurrent oncological diseases
* need for chronic use of medication that may affect BP levels
* pregnancy
* history of narcolepsy or restless leg syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
drop in blood pressure | two years

CONTACTS AND LOCATIONS:
Overall Officials: Sophia E Schiza, MD, PhD, Study Chair — University of Crete
Locations (1):
- Sleep Disorders Center, Department of Thoracic Medicine, University of Crete,, Heraklion, Greece